CLINICAL TRIAL: NCT02969603
Title: Evaluation of Leg Muscular Activity Using Magnetic Resonance Imaging and 11C-acetate Positron Tomography (PET/MRI). Pilot Study
Brief Title: Evaluation of Leg Muscular Activity Using MRI and 11C-acetate PET/MRI. Pilot Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Osman Ratib (Other)
Responsible Party: Sponsor-Investigator, Osman Ratib, Dr., University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013DR2115
Record Dates: First submitted 2016-04-14; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: PET/MRI; muscular activity; 11C-acetate
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers- MRI (Other): MRI scan for morphological assessment of muscle structures and anatomy
  Interventions: Other: Magnetic Resonance Imaging
- Healthy Volunteers- PET/MRI (Other): The volunteers will undergo a combined [11C]acetate PET/MRI scan
  Interventions: Other: Magnetic Resonance combined with Positron Emission Tomography

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Magnetic Resonance Imaging as reference
  Arms: Healthy volunteers- MRI
Other: Magnetic Resonance combined with Positron Emission Tomography — Comparison with MRI only, to assess muscular activity, creation of anatomic images of muscle activity and resolution of metabolic activity distribution within exercising skeletal muscle
  Arms: Healthy Volunteers- PET/MRI

SUMMARY:
The present study is conceived as a pilot study aimed to determine the efficiency of the newly available Positron Emission Tomography (PET) - Magnetic Resonance Imaging (MRI) hybrid scan technique for muscular activity evaluation, creation of anatomic images of muscle activity and resolution of metabolic activity distribution within exercising skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

MRI exam inclusion criteria

* Male volunteer aged in the range 18 to 35 years.
* Acceptance of the research protocol: signature of the informed consent form after oral and written information about the protocol through the patient information document.
* Volunteers that could undergo 1h15 to 1h30 immobilization (MRI exam duration in time).

PET/MRI exam inclusion criteria

* Male volunteer aged in the range 18 to 35 years.
* Acceptance of the research protocol: signature of the informed consent form after oral and written information about the protocol through the patient information document.
* Volunteers that could undergo 1.5 to 2.0 hours immobilization (PET/MRI exam duration in time).
* Volunteers should practice regular physical activity, defined as 50 min per day (in a single session), 2 days per week of physical activity as a minimum (no maximum is fixed).

Exclusion criteria MRI exam exclusion criteria

* Pre-existing neurological or muscular lesions on the legs.
* Co morbidities impeding on the protocol comprehension or fulfilment.
* Illnesses that do not allow to lay down on an examination table.
* Pacemaker holder.
* Metal implants that would preclude MRI imaging
* Claustrophobia: Subjects will be questioned about possible discomfort with being in an enclosed space (e.g., MRI scanner). Those who report such problems will be excluded.

PET/MRI exam exclusion criteria

* Medical radiation exposure within the last five years (normal population should not be exposed to medical radiation higher or equal to 1 mSv per year).
* Pre-existing neurological or muscular lesions on the legs.
* Co morbidities impeding on the protocol comprehension or fulfilment.
* Illnesses that do not allow to lay down on an examination table.
* Pacemaker holder.
* Metal implants that would preclude MRI imaging
* Claustrophobia: Subjects will be questioned about possible discomfort with being in an enclosed space (e.g., MRI scanner). Those who report such problems will be excluded.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of musculoskeletal systems in motion | though study completion, an average of 2 years
  an informatic visualization tool of muscles implied in leg flexion/extension combining PET and MR infomation
Distribution of acetate metabolism during exercise skeletal muscle | though study completion, an average of 2 years
  11C-acetate uptake (SUV and SUVratio with resting muscles) in contracting muscle, measured using muscle segmentation from MRI images

SECONDARY OUTCOMES:
Measurement of the in vivo function of the muscle | though study completion, an average of 2 years
  correlation between 11C-acetate uptake and contractile force measures (weight and duration of exercise)

CONTACTS AND LOCATIONS:
Overall Officials: Osman Ratib, Pr., Principal Investigator — University Hospital, Geneva
Locations (1):
- Service de Medecine Nucléaire et Imagerie moléculaire- HUG, Geneva, Switzerland